CLINICAL TRIAL: NCT06205784
Title: Prehabilitative Exercise - Can the Physiological Consequences of Immobilization be Prevented?
Brief Title: Prehabilitative Exercise Prior to Immobilization
Acronym: PREHAB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Casper Soendenbroe, Postdoc, Bispebjerg Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: BBH164
Record Dates: First submitted 2023-12-19; First posted 2024-01-16 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Sarcopenia; Skeletal Muscle Atrophy; Disuse Atrophy
MeSH Terms: conditions — Sarcopenia; Muscular Atrophy; Muscular Disorders, Atrophic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Prehab (Experimental)
  Interventions: Other: Prehabilitative exercise
- NoTrain (No Intervention)

INTERVENTIONS:
Other: Prehabilitative exercise — 3-4 weeks of heavy resistance exercise
  Arms: Prehab

SUMMARY:
This is a 10-week human study involving 24 younger (20-35 y) and 24 older (65-85 y) healthy individuals. All participants will undergo unilateral immobilization of a knee for 7-10 days, followed by 4 weeks of heavy resistance exercise training (HReT). Half of the participants (12 younger and 12 older) will also undergo 4 weeks HReT prior to the immobilization. Prehabilitative exercise may confer protective effects on subsequent immobilization, and the various underlying mechanisms involved

ELIGIBILITY:
Inclusion Criteria:

* Age: Between 20-35 years old or between 65-85 years old.
* BMI: Between 18.5 and 35 kg/m2.
* Healthy and well, with normal dietary habits (not vegan).

Exclusion Criteria:

* More than one muscle biopsy previously taken from both vastus lateralis muscles.
* Smoking.
* Pregnancy.
* Past or present substance or alcohol abuse.
* Medical/surgical conditions that are assessed to affect protein synthesis or the participant's involvement in the trial.
* Knee pain that could affect the completion of the training intervention.
* High intake of supplements that increase the risk of bleeding during muscle biopsy (such as fish oil and ginger).
* Participation in regular strength training within the past year.
* Regular participation in structured sports.
* Current use of blood-thinning medication.
* Previous participation in trials involving oral intake of heavy water.
* Metal in the body preventing MRI scanning.
* For the older group, not having gone through menopause, and for the younger group, not having a regular menstrual cycle.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2024-01-06 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Quadriceps cross-sectional area | From pre (week 0) to post immobilization (week 5)
  Quadriceps cross-sectional area measured by MRI

SECONDARY OUTCOMES:
Muscle fiber size | From pre (week 0) to post immobilization (week 5) and post retraining (week 10)
  Muscle fiber size assessed by histochemical stainings
Denervated muscle fibers | From pre (week 0) to post immobilization (week 5) and post retraining (week 10)
  Assessment denervated fibers using histochemical stainings
Muscle protein synthesis | From pre immobilization (week 4) to post immobilization (week 5)
  Muscle protein synthesis assessed using deuterium (heavy water)
Muscle gene expression | From pre (week 0) to post immobilization (week 5) and post retraining (week 10)
  Muscle gene expression assessed by RNA sequencing
Brain structure | From pre (week 0) to post immobilization (week 5) and post retraining (week 10)
  Brain structure measured by MRI
Brain function | From pre (week 0) to post immobilization (week 5) and post retraining (week 10)
  Brain function measured by MRI
Tendon structure | From pre (week 0) to post immobilization (week 5)
  Tendon structure measured by MRI
Tendon ultrastructure | From pre immobilization (week 4) to post immobilization (week 5)
  Tendon tissue analysed by molecular analyses
Lean-body mass | From pre (week 0) to post immobilization (week 5) and post retraining (week 10)
  Whole-body and thigh lean-body mass assessed using DEXA-scans
Muscle strength | From pre (week 0) to post immobilization (week 5) and post retraining (week 10)
  Muscle strength during knee extension assessed using isokinetic and isometric dynamometers
Balance | From pre (week 0) to post immobilization (week 5) and post retraining (week 10)
  One-legged balanced assessed using a force platform
Force variability | From pre (week 0) to post immobilization (week 5) and post retraining (week 10)
  Force variability during knee extension assessed using submaximal isometric contractions

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Sports Medicine Copenhagen, Copenhagen, Capital Region, Denmark

IPD SHARING:
Plan to Share IPD: Undecided